CLINICAL TRIAL: NCT06470412
Title: Personalized Management of Autoimmune Diseases With AI-Guided (GenAIS TM) Dietary Supplementation: A Randomized Controlled Study
Brief Title: Personalized Management of Autoimmune Diseases With AI-Guided (GenAIS TM) Dietary Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Triangel Scientific (Industry); Center of New Medical Technologies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW015
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-06

CONDITIONS: Autoimmune Diseases
Keywords: AI-guided dietary supplementation; Genetic profiling; Metabolic profiling; Disease reduction
MeSH Terms: conditions — Autoimmune Diseases | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Other: Control group
- AI-Guided Group (Experimental)
  Interventions: Other: AI-Guided Group

INTERVENTIONS:
Other: Control group — Participants receive supplement prescriptions from a physician based on current standard practices, which include biochemical markers, genetic data, and metabolic profiles.
  Arms: Control Group
Other: AI-Guided Group — Participants receive supplement prescriptions determined by GenAIS, an AI system which considers genetic data, metabolic profiles, biochemical markers, and patient history.
  Arms: AI-Guided Group

SUMMARY:
The study "Personalized Management of Autoimmune Diseases with AI-Guided (GenAIS TM) Dietary Supplementation" investigated the effectiveness of AI-guided dietary supplement (DS) prescriptions compared to standard physician-guided prescriptions in managing autoimmune diseases. This 6-month randomized controlled trial included 160 participants with conditions like rheumatoid arthritis, lupus, and multiple sclerosis. Participants were divided into two groups: one received DS based on physician judgment, and the other based on GenAIS AI system analysis. Primary outcomes focused on changes in disease activity, while secondary outcomes included quality of life, metabolic markers, and DS adherence. Data collection involved genetic, metabolic, and clinical profiling, with ethical considerations ensuring participant confidentiality and informed consent

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with an autoimmune disease (e.g., rheumatoid arthritis, lupus, multiple sclerosis) according to established clinical criteria.
* Moderate to severe disease activity as indicated by standardized measures (e.g., DAS28 for rheumatoid arthritis, SLEDAI for lupus).
* Stable on existing autoimmune medication regimen for at least 3 months prior to the study.
* Willingness to provide genetic and metabolic data.
* Written informed consent.

Exclusion Criteria:

* Current or past history of severe psychiatric conditions or other severe chronic diseases.
* Significant medical conditions like severe renal, hepatic, or cardiovascular diseases that may interfere with the study outcomes.
* Use of dietary supplements that affect immune function within the last 3 months.
* Pregnancy or breastfeeding.
* Recent changes in autoimmune medication within the last 3 months.
* Participation in another clinical trial within the last 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
The percent change in disease activity scores for the AI-Guided group compared with the Control group | 6 months
  Systemic Lupus Erythematosus Disease Activity Index, which has a score range from 0 to 105, to measure disease activity in participants with lupus.
  Disease Activity Score 28 (DAS28), which has a score range from 0 to 10, to measure disease activity in participants with rheumatoid arthritis.

SECONDARY OUTCOMES:
Percent change in specific symptoms of autoimmune disease | 6 months
Percent change in high-sensitivity C-reactive protein | 6 months
Percent change in body weight and body mass index | 6 months
Incidence of adverse effects related to dietary supplements. | 6 months
Number Participant adherence to the prescribed dietary supplements regimen | 6 months
Changes in quality of life score Short Form-36 | 6 months
  Short Form-36 Health Survey, which has a score range from 0 to 100, to measure the quality of life in participants, with higher scores indicating better health and well-being.
Changes in quality of life score World Health Organization Quality of Life - BREF | 6 months
  World Health Organization Quality of Life - BREF, which has a score range from 0 to 100, to measure the quality of life in participants, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia